CLINICAL TRIAL: NCT02710630
Title: Relative Bioavailability of Dabigatran After Single Oral Administration of Five Different Tablet Formulations of Dabigatran Etexilate Compared to Commercial Capsule Formulation in Healthy Male Subjects (an Open-label, Randomised, Single-dose, Six-period, Five-sequence Crossover Study)
Brief Title: Bioavailability Study of Five Tablet Formulations of Dabigatran Etexilate Compared to Commercial Capsule Formulation in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.246
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran

ARMS (6):
- Dabigatran etexilate capsule (Active Comparator)
  Interventions: Drug: Dabigatran etexilate capsule
- Dabigatran etexilate tablet A1 (Experimental)
  Interventions: Drug: Dabigatran etexilate tablet A1
- Dabigatran etexilate tablet B1 (Experimental)
  Interventions: Drug: Dabigatran etexilate tablet B1
- Dabigatran etexilate tablet C1 (Experimental)
  Interventions: Drug: Dabigatran etexilate tablet C1
- Dabigatran etexilate tablet D1 (Experimental)
  Interventions: Drug: Dabigatran etexilate tablet D1
- Dabigatran etexilate tablet E1 (Experimental)
  Interventions: Drug: Dabigatran etexilate tablet E1

INTERVENTIONS:
Drug: Dabigatran etexilate tablet E1
  Arms: Dabigatran etexilate tablet E1
Drug: Dabigatran etexilate tablet D1
  Arms: Dabigatran etexilate tablet D1
Drug: Dabigatran etexilate tablet C1
  Arms: Dabigatran etexilate tablet C1
Drug: Dabigatran etexilate tablet B1
  Arms: Dabigatran etexilate tablet B1
Drug: Dabigatran etexilate tablet A1
  Arms: Dabigatran etexilate tablet A1
Drug: Dabigatran etexilate capsule
  Arms: Dabigatran etexilate capsule

SUMMARY:
The primary objective of this trial is to investigate the relative bioavailability of five different tablet formulations of Dabigatran Etexilate, Formulation A1, Formulation B1, Formulation C1, Formulation D1, and Formulation E1, compared to commercial capsule formulation of Dabigatran Etexilate.

The secondary objective is to evaluate and compare several pharmacokinetic parameters between the treatments.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (blood pressure [BP], pulse rate [PR]), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age >=20 and <=35 years old
* Body mass index (BMI) >=18.0 and <=25.0 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

* Any finding in the medical examination (including BP, Pulse Rate, or ECG) deviating from normal and judged as clinically relevant by the investigator at screening
* Measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm at screening
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any relevant bleeding history considered by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* Any history or evidence of blood dyscrasia, haemorrhagic diathesis, severe thrombocytopenia, cerebrovascular haemorrhage, bleeding tendencies associated with active ulceration or overt bleeding of gastrointestinal, respiratory or genitourinary tract or any disease or condition with haemorrhagic tendencies
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Any evidence of a concomitant disease considered as clinically relevant by the investigator
* Intake of drugs with a long half-life (more than 24 hours) within 30 days or less than 10 half-lives of the respective drug prior to administration of trial medication
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial
* Intake of medication, which influences the blood clotting, e.g., acetylsalicylic acid, coumarin etc. within 10 days prior to trial medication
* Participation in another trial where an investigational drug has been administered within 4 months or 5 half-lives (whichever is greater) prior to planned administration of trial medication
* Planned surgeries within four weeks following the end-of study examination
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking during in-house confinement at the trial site
* Alcohol abuse (consumption of more than 30 g per day: e.g., 750 mL of beer, 1.5 gous [equivalent to 270 mL] of Sake)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* Subject assessed as unsuitable for inclusion by the investigator because of, for instance, being considered not able to understand and comply with study requirements, or having a condition that would not allow safe participation in the study

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2016-05-11 (Actual); Study Completion 2016-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Ref-A1-B1-C1-D1-E1: All subjects were treated with the reference treatment (Ref), Dabigatran Etexilate (BIBR 1048) commercial capsule formulation, 110 mg orally (one day, single dose) with 200 mL of water after an overnight fast of at least 10 hours in period 1, followed by one of the 5 investigational treatment in the following sequence, i.e., test formulation Dabigatran Etexilate tablet formulations in the sequence Test Formulation A1 (TF-A1) in period 2, followed by Test Formulation B1 (TF-B1) in period 3, followed by Test Formulation C1 (TF-C1) in period 4, followed by Test Formulation D1 (TF-D1) in period 5, followed by Test Formulation E1 (TF-E1) in period 6, 110 mg orally (one day, single dose) with 200 mL of water after an overnight fast of at least 10 hours.
  A washout period of at least 4 days was set following the drug administration in each period.
- Ref-B1-C1-D1-E1-A1: All subjects were treated with the reference treatment (Ref), Dabigatran Etexilate (BIBR 1048) commercial capsule formulation, 110 mg orally (one day, single dose) with 200 mL of water after an overnight fast of at least 10 hours in period 1, followed by one of the 5 investigational treatment in the following sequence, i.e., test formulation Dabigatran Etexilate tablet formulations in the sequence Test Formulation B1 (TF-B1) in period 2, followed by Test Formulation C1 (TF-C1) in period 3, followed by Test Formulation D1 (TF-D1) in period 4, followed by Test Formulation E1 (TF-E1) in period 5, followed by Test Formulation A1 (TF-A1) in period 6, 110 mg orally (one day, single dose) with 200 mL of water after an overnight fast of at least 10 hours.
  A washout period of at least 4 days was set following the drug administration in each period.
- Ref-C1-D1-E1-A1-B1: All subjects were treated with the reference treatment (Ref), Dabigatran Etexilate (BIBR 1048) commercial capsule formulation, 110 mg orally (one day, single dose) with 200 mL of water after an overnight fast of at least 10 hours in period 1, followed by one of the 5 investigational treatment in the following sequence, i.e., test formulation Dabigatran Etexilate tablet formulations in the sequence Test Formulation C1 (TF-C1) in period 2, followed by Test Formulation D1 (TF-D1) in period 3, followed by Test Formulation E1 (TF-E1) in period 4, followed by Test Formulation A1 (TF-A1) in period 5, followed by Test Formulation B1 (TF-B1) in period 6, 110 mg orally (one day, single dose) with 200 mL of water after an overnight fast of at least 10 hours.
  A washout period of at least 4 days was set following the drug administration in each period.
- Ref-D1-E1-A1-B1-C1: All subjects were treated with the reference treatment (Ref), Dabigatran Etexilate (BIBR 1048) commercial capsule formulation, 110 mg orally (one day, single dose) with 200 mL of water after an overnight fast of at least 10 hours in period 1, followed by one of the 5 investigational treatment in the following sequence, i.e., test formulation Dabigatran Etexilate tablet formulations in the sequence Test Formulation D1 (TF-D1) in period 2, followed by Test Formulation E1 (TF-E1) in period 3, followed by Test Formulation A1 (TF-A1) in period 4, followed by Test Formulation B1 (TF-B1) in period 5, followed by Test Formulation C1 (TF-C1) in period 6, 110 mg orally (one day, single dose) with 200 mL of water after an overnight fast of at least 10 hours.
  A washout period of at least 4 days was set following the drug administration in each period.
- Ref-E1-A1-B1-C1-D1: All subjects were treated with the reference treatment (Ref), Dabigatran Etexilate (BIBR 1048) commercial capsule formulation, 110 mg orally (one day, single dose) with 200 mL of water after an overnight fast of at least 10 hours in period 1, followed by one of the 5 investigational treatment in the following sequence, i.e., test formulation Dabigatran Etexilate tablet formulations in the sequence Test Formulation E1 (TF-E1) in period 2, followed by Test Formulation A1 (TF-A1) in period 3, followed by Test Formulation B1 (TF-B1) in period 4, followed by Test Formulation C1 (TF-C1) in period 5, followed by Test Formulation D1 (TF-D1) in period 6, 110 mg orally (one day, single dose) with 200 mL of water after an overnight fast of at least 10 hours.
  A washout period of at least 4 days was set following the drug administration in each period.
Period: Period 1
Arm/Group | Ref-A1-B1-C1-D1-E1 | Ref-B1-C1-D1-E1-A1 | Ref-C1-D1-E1-A1-B1 | Ref-D1-E1-A1-B1-C1 | Ref-E1-A1-B1-C1-D1
Started | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Ref-A1-B1-C1-D1-E1 | Ref-B1-C1-D1-E1-A1 | Ref-C1-D1-E1-A1-B1 | Ref-D1-E1-A1-B1-C1 | Ref-E1-A1-B1-C1-D1
Started | 7 | 7 | 7 | 7 | 7
Not Treated | 1 | 0 | 0 | 0 | 0
Completed | 7 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Ref-A1-B1-C1-D1-E1 | Ref-B1-C1-D1-E1-A1 | Ref-C1-D1-E1-A1-B1 | Ref-D1-E1-A1-B1-C1 | Ref-E1-A1-B1-C1-D1
Started | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Ref-A1-B1-C1-D1-E1 | Ref-B1-C1-D1-E1-A1 | Ref-C1-D1-E1-A1-B1 | Ref-D1-E1-A1-B1-C1 | Ref-E1-A1-B1-C1-D1
Started | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Ref-A1-B1-C1-D1-E1 | Ref-B1-C1-D1-E1-A1 | Ref-C1-D1-E1-A1-B1 | Ref-D1-E1-A1-B1-C1 | Ref-E1-A1-B1-C1-D1
Started | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 6
Arm/Group | Ref-A1-B1-C1-D1-E1 | Ref-B1-C1-D1-E1-A1 | Ref-C1-D1-E1-A1-B1 | Ref-D1-E1-A1-B1-C1 | Ref-E1-A1-B1-C1-D1
Started | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This set included all subjects that were dispensed study drug and were documented to have taken at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ref-A1-B1-C1-D1-E1 | Ref-B1-C1-D1-E1-A1 | Ref-C1-D1-E1-A1-B1 | Ref-D1-E1-A1-B1-C1 | Ref-E1-A1-B1-C1-D1 | Total
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.9 (2.4) | 28.1 (3.4) | 27.3 (3.4) | 29.1 (3.6) | 27.4 (3.4) | 27.8 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 7 | 7 | 7 | 7 | 7 | 35

OUTCOME MEASURES:

1. Primary Outcome: AUC0-tz (Area Under the Concentration-time Curve of Free Dabigatran in Plasma Over the Time Interval From 0 to the Time of the Last Quantifiable Data Point)
Description: This outcome measure presents area under the concentration-time curve of free Dabigatran in plasma over the time interval from 0 to the time of the last quantifiable data point.
Time Frame: 1:00 [hour (h): minute] before drug administration and 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 12:00h, 24:00h, 36:00h, 48:00h after drug administration.
Population: The PharmacoKinetic (PK) parameter analysis Set (PKS): This analysis set included all subjects of the treated set who provided at least one primary or secondary PK parameter. Thus, a subject was included in the PKS, even if the subject contributed only one PK parameter value for one period to the statistical assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Dabigatran Etexilate Capsule: Ref: The subjects received Dabigatran Etexilate (Reference) capsule formulation (commercial formulation) 110 mg orally (one day, single dose) with 200 mL of water after an overnight fast of at least 10 hours.
- Dabigatran Etexilate Tablet: A1: The subjects received Dabigatran Etexilate (Test) tablet formulation (A1), 110 mg orally (one day, single dose) with 200 mL of water after an overnight fast of at least 10 hours.
- Dabigatran Etexilate Tablet: B1: The subjects received Dabigatran Etexilate (Test) tablet formulation (B1), 110 mg orally (one day single dose) with 200 mL of water after an overnight fast of at least 10 hours.
- Dabigatran Etexilate Tablet: C1: The subjects received Dabigatran Etexilate (Test) tablet formulation (C1), 110 mg orally (one day single dose) with 200 mL of water after an overnight fast of at least 10 hours.
- Dabigatran Etexilate Tablet: D1: The subjects received Dabigatran Etexilate (Test) tablet formulation (D1), 110 mg orally (one day single dose) with 200 mL of water after an overnight fast of at least 10 hours.
- Dabigatran Etexilate Tablet: E1: The subjects received Dabigatran Etexilate (Test) tablet formulation (E1), 110 mg orally (one day single dose) with 200 mL of water after an overnight fast of at least 10 hours.
Arm/Group | Dabigatran Etexilate Capsule: Ref | Dabigatran Etexilate Tablet: A1 | Dabigatran Etexilate Tablet: B1 | Dabigatran Etexilate Tablet: C1 | Dabigatran Etexilate Tablet: D1 | Dabigatran Etexilate Tablet: E1
Number analyzed (Participants) | 35 | 34 | 35 | 35 | 35 | 35
ng*h/mL | 600 (51.8) | 714 (42.1) | 318 (327) | 354 (96.6) | 649 (78.6) | 661 (54.8)
Statistical Analysis 1: Comparison: Dabigatran Etexilate Tablet: A1; Test type: Superiority or Other; Ratio [Test/Reference] = 119.33, 90% CI 2-sided [101.838 to 139.834], Standard Deviation 40.4 — The adjusted geometric mean (gMean) ratio [%] calculated as Dabigatran Etexilate Tablet: A1/Dabigatran Etexilate Capsule: Ref. Standard deviation is actually intra-individual geometric coefficient of variation (gCV) [%]
Statistical Analysis 2: Comparison: Dabigatran Etexilate Tablet: B1; Test type: Superiority or Other; Ratio [Test/Reference] = 52.97, 90% CI 2-sided [33.341 to 84.158], Standard Deviation 168.9 — The adjusted geometric mean (gMean) ratio [%] calculated as Dabigatran Etexilate Tablet: B1/Dabigatran Etexilate Capsule: Ref. Standard deviation is actually intra-individual geometric coefficient of variation (gCV) [%]
Statistical Analysis 3: Comparison: Dabigatran Etexilate Tablet: C1; Test type: Superiority or Other; Ratio [Test/Reference] = 59.01, 90% CI 2-sided [45.255 to 76.955], Standard Deviation 73.4 — The adjusted geometric mean (gMean) ratio [%] calculated as Dabigatran Etexilate Tablet: C1/Dabigatran Etexilate Capsule: Ref. Standard deviation is actually intra-individual geometric coefficient of variation (gCV) [%]
Statistical Analysis 4: Comparison: Dabigatran Etexilate Tablet: D1; Test type: Superiority or Other; Ratio [Test/Reference] = 108.21, 90% CI 2-sided [87.698 to 133.530], Standard Deviation 55.7 — The adjusted geometric mean (gMean) ratio [%] calculated as Dabigatran Etexilate Tablet: D1/Dabigatran Etexilate Capsule: Ref. Standard deviation is actually intra-individual geometric coefficient of variation (gCV) [%]
Statistical Analysis 5: Comparison: Dabigatran Etexilate Tablet: E1; Test type: Superiority or Other; Ratio = 110.21, 90% CI 2-sided [93.939 to 129.297], Standard Deviation 41.1 — The adjusted geometric mean (gMean) ratio [%] calculated as Dabigatran Etexilate Tablet: E1/Dabigatran Etexilate Capsule: Ref. Standard deviation is actually intra-individual geometric coefficient of variation (gCV) [%]

2. Primary Outcome: Cmax (Maximum Concentration of Free Dabigatran)
Description: This outcome measure presents maximum concentration of analyte in plasma (Cmax).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabigatran Etexilate Capsule: Ref | Dabigatran Etexilate Tablet: A1 | Dabigatran Etexilate Tablet: B1 | Dabigatran Etexilate Tablet: C1 | Dabigatran Etexilate Tablet: D1 | Dabigatran Etexilate Tablet: E1
Number analyzed (Participants) | 35 | 34 | 35 | 35 | 35 | 35
ng/mL | 73.5 (60.0) | 86.8 (39.3) | 42.3 (213) | 45.5 (81.5) | 79.6 (73.5) | 79.2 (52.7)
Statistical Analysis 1: Comparison: Dabigatran Etexilate Tablet: A1; Test type: Superiority or Other; Ratio [Test/Reference] = 118.31, 90% CI 2-sided [99.569 to 140.579], Standard Deviation 44.2 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Dabigatran Etexilate Tablet: B1; Test type: Superiority or Other; Ratio [Test/Reference] = 57.49, 90% CI 2-sided [38.502 to 85.837], Standard Deviation 132.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Dabigatran Etexilate Tablet: C1; Test type: Superiority or Other; Ratio [Test/Reference] = 61.94, 90% CI 2-sided [48.130 to 79.720], Standard Deviation 69.0 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Dabigatran Etexilate Tablet: D1; Test type: Superiority or Other; Ratio [Test/Reference] = 108.26, 90% CI 2-sided [87.704 to 133.629], Standard Deviation 55.8 — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Dabigatran Etexilate Tablet: E1; Test type: Superiority or Other; Ratio [Test/Reference] = 107.76, 90% CI 2-sided [91.238 to 127.281], Standard Deviation 43.0 — [estimate comment as in outcome 1, analysis 5]

3. Secondary Outcome: AUC0-infinity (Area Under the Concentration-time Curve of Free Dabigatran in Plasma Over the Time Interval From 0 Extrapolated to Infinity) (if Applicable)
Description: This outcome measure presents area under the concentration-time curve of free Dabigatran in plasma over the time interval from 0 extrapolated to infinity)(if applicable).
Time Frame: as for outcome 1
Population: The PharmacoKinetic (PK) parameter analysis Set (PKS): Included all subjects of the treated set who provided at least one primary or secondary PK parameter.
  PK Set 2 (PKS2): Included all subjects in the PKS who had evaluable PK variable of the reference treatment and at least one of the 5 test treatments.
  PKS2 was used for statistical analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dabigatran Etexilate Capsule: Ref | Dabigatran Etexilate Tablet: A1 | Dabigatran Etexilate Tablet: B1 | Dabigatran Etexilate Tablet: C1 | Dabigatran Etexilate Tablet: D1 | Dabigatran Etexilate Tablet: E1
Number analyzed (Participants) | 35 | 34 | 31 | 32 | 34 | 35
ng*h/mL | 623 (49.0) | 735 (40.2) | 544 (71.9) | 444 (60.3) | 725 (53.0) | 684 (51.9)
Statistical Analysis 1: Comparison: Dabigatran Etexilate Tablet: A1; Test type: Superiority or Other; Ratio [Test/Reference] = 118.26, 90% CI 2-sided [101.627 to 137.621], Standard Deviation 38.5 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Dabigatran Etexilate Tablet: B1; Test type: Superiority or Other; Ratio [Test/Reference] = 87.26, 90% CI 2-sided [69.404 to 109.722], Standard Deviation 60.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Dabigatran Etexilate Tablet: C1; Test type: Superiority or Other; Ratio [Test/Reference] = 71.40, 90% CI 2-sided [58.828 to 86.648], Standard Deviation 49.2 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Dabigatran Etexilate Tablet: D1; Test type: Superiority or Other; Ratio [Test/Reference] = 116.67, 90% CI 2-sided [100.516 to 135.410], Standard Deviation 37.7 — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Dabigatran Etexilate Tablet: E1; Test type: Superiority or Other; Ratio [Test/Reference] = 109.85, 90% CI 2-sided [94.452 to 127.750], Standard Deviation 38.7 — [estimate comment as in outcome 1, analysis 5]

4. Secondary Outcome: AUC0-tz (Area Under the Concentration-time Curve of Total Dabigatran in Plasma Over the Time Interval From 0 to the Time of the Last Quantifiable Data Point)
Description: This outcome measure presents area under the concentration-time curve of total Dabigatran in plasma over the time interval from 0 to the time of the last quantifiable data point.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dabigatran Etexilate Capsule: Ref | Dabigatran Etexilate Tablet: A1 | Dabigatran Etexilate Tablet: B1 | Dabigatran Etexilate Tablet: C1 | Dabigatran Etexilate Tablet: D1 | Dabigatran Etexilate Tablet: E1
Number analyzed (Participants) | 35 | 34 | 35 | 35 | 35 | 35
ng*h/mL | 726 (52.9) | 838 (41.1) | 366 (341) | 412 (97.1) | 777 (74.9) | 778 (53.6)
Statistical Analysis 1: Comparison: Dabigatran Etexilate Tablet: A1; Test type: Superiority or Other; Ratio [Test/Reference] = 115.69, 90% CI 2-sided [98.783 to 135.491], Standard Deviation 40.2 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Dabigatran Etexilate Tablet: B1; Test type: Superiority or Other; Ratio [Test/Reference] = 50.43, 90% CI 2-sided [31.519 to 80.689], Standard Deviation 173.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Dabigatran Etexilate Tablet: C1; Test type: Superiority or Other; Ratio [Test/Reference] = 56.71, 90% CI 2-sided [43.388 to 74.122], Standard Deviation 74.2 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Dabigatran Etexilate Tablet: D1; Test type: Superiority or Other; Ratio [Test/Reference] = 106.99, 90% CI 2-sided [87.554 to 130.732], Standard Deviation 52.8 — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Dabigatran Etexilate Tablet: E1; Test type: Superiority or Other; Ratio [Test/Reference] = 107.07, 90% CI 2-sided [91.399 to 125.432], Standard Deviation 40.7 — [estimate comment as in outcome 1, analysis 5]

5. Secondary Outcome: Cmax (Maximum Plasma Concentration of Total Dabigatran)
Description: This outcome measure presents maximum concentration of analyte in plasma (Cmax).
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabigatran Etexilate Capsule: Ref | Dabigatran Etexilate Tablet: A1 | Dabigatran Etexilate Tablet: B1 | Dabigatran Etexilate Tablet: C1 | Dabigatran Etexilate Tablet: D1 | Dabigatran Etexilate Tablet: E1
Number analyzed (Participants) | 35 | 34 | 35 | 35 | 35 | 35
ng/mL | 88.6 (62.0) | 102 (39.0) | 47.9 (227) | 52.2 (83.6) | 94.2 (75.7) | 91.9 (54.1)
Statistical Analysis 1: Comparison: Dabigatran Etexilate Tablet: A1; Test type: Superiority or Other; Ratio [Test/Reference] = 115.39, 90% CI 2-sided [96.740 to 137.644], Standard Deviation 45.3 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Dabigatran Etexilate Tablet: B1; Test type: Superiority or Other; Ratio [Test/Reference] = 54.12, 90% CI 2-sided [35.818 to 81.774], Standard Deviation 138.6 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Dabigatran Etexilate Tablet: C1; Test type: Superiority or Other; Ratio [Test/Reference] = 58.96, 90% CI 2-sided [45.489 to 76.431], Standard Deviation 71.4 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Dabigatran Etexilate Tablet: D1; Test type: Superiority or Other; Ratio [Test/Reference] = 106.38, 90% CI 2-sided [85.846 to 131.836], Standard Deviation 57.0 — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Dabigatran Etexilate Tablet: E1; Test type: Superiority or Other; Ratio [Test/Reference] = 103.73, 90% CI 2-sided [87.740 to 122.628], Standard Deviation 43.3 — [estimate comment as in outcome 1, analysis 5]

6. Secondary Outcome: AUC0-infinity (Area Under the Concentration-time Curve of Total Dabigatran in Plasma Over the Time Interval From 0 Extrapolated to Infinity) (if Applicable)
Description: This outcome measure presents area under the concentration-time curve of total Dabigatran in plasma over the time interval from 0 extrapolated to infinity)(if applicable).
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dabigatran Etexilate Capsule: Ref | Dabigatran Etexilate Tablet: A1 | Dabigatran Etexilate Tablet: B1 | Dabigatran Etexilate Tablet: C1 | Dabigatran Etexilate Tablet: D1 | Dabigatran Etexilate Tablet: E1
Number analyzed (Participants) | 35 | 34 | 31 | 32 | 35 | 35
ng*h/mL | 750 (50.5) | 863 (39.1) | 628 (75.6) | 515 (60.1) | 804 (70.1) | 800 (51.9)
Statistical Analysis 1: Comparison: Dabigatran Etexilate Tablet: A1; Test type: Superiority or Other; Ratio [Test/Reference] = 115.27, 90% CI 2-sided [99.063 to 134.130], Standard Deviation 38.4 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Dabigatran Etexilate Tablet: B1; Test type: Superiority or Other; Ratio [Test/Reference] = 83.73, 90% CI 2-sided [66.033 to 106.163], Standard Deviation 62.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Dabigatran Etexilate Tablet: C1; Test type: Superiority or Other; Ratio [Test/Reference] = 68.77, 90% CI 2-sided [56.452 to 83.782], Standard Deviation 50.3 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Dabigatran Etexilate Tablet: D1; Test type: Superiority or Other; Ratio [Test/Reference] = 107.13, 90% CI 2-sided [88.616 to 129.510], Standard Deviation 49.6 — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Dabigatran Etexilate Tablet: E1; Test type: Superiority or Other; Ratio [Test/Reference] = 106.64, 90% CI 2-sided [91.625 to 124.114], Standard Deviation 38.9 — [estimate comment as in outcome 1, analysis 5]

ADVERSE EVENTS:
Time Frame: From first drug administration until 1 day after last drug administration, up to 81 days.
Arm/Group | Dabigatran Etexilate Capsule: Ref | Dabigatran Etexilate Tablet: A1 | Dabigatran Etexilate Tablet: B1 | Dabigatran Etexilate Tablet: C1 | Dabigatran Etexilate Tablet: D1 | Dabigatran Etexilate Tablet: E1
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34 | 0/35 | 0/35 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/34 | 0/35 | 0/35 | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.